CLINICAL TRIAL: NCT02935595
Title: A Systematic Investigation of Neurophysiological Correlates of Low Dose Intravenous Ketamine in Treatment Resistant Depression Patients
Brief Title: Low Dose Intravenous Ketamine in Treatment Resistant Depression Patients
Acronym: ketamine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Sudhakar Selvaraj, MBBS., DPhil (Oxon)., MRCPsych, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-16-0705
Record Dates: First submitted 2016-10-12; First posted 2016-10-17 (Estimated); Results first posted 2020-08-31 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Open-label
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ketamine (Experimental): Slow infusions of ketamine will take place over a time period of 40 minutes.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Ketamine Hydrochloride Injection
  Other Names: Ketamine Hydrochloride

SUMMARY:
The primary goal of the project is to study the effect of Ketamine on cortical neurophysiological function in TRD patients. The proposal employs robust and non-invasive neurophysiological techniques TMS and EEG to investigate the cortical excitability and oscillatory activity in patients with treatment resistant depression.

DETAILED DESCRIPTION:
The primary goal of the project is to study the effect of Ketamine on cortical neurophysiological function in Treatment Resistant Depression(TRD) patients. There are three key preclinical findings regarding Ketamine antidepressant effects that motivate the current study: a) low dose Ketamine causes early increase in glutamate neurotransmission; b) Ketamine initiates synaptic plasticity; c) ketamine infusion leads to rapid improvement in depression symptoms. The proposal essentially employs robust and non-invasive neurophysiological techniques, Auditory Steady State Response(ASSR)-gamma oscillatory response and Transcranial Magnetic Stimulation(TMS) cortical excitability to investigate the above findings in patients with treatment resistant depression.

Study:

Ketamine Infusion:

We will employ an open-label study in which the infusion session, the enrolled TRD patients will receive low dose Ketamine (0.5 mg/kg) over 40 minutes.

Cortical Excitability:

TMS stimulation will be applied to the corresponding region of the contralateral primary motor cortex to determine motor threshold and to examine the motor cortical excitability measures after Ketamine. The optimal coil position will be determined by moving the TMS coil in 1-cm increments over the motor cortical area while delivering single or paired magnetic pulses and by observing maximal contraction of the contralateral abductor pollicis brevis (APB). Electromyography readings will be obtained from the APB muscle. TMS stimulation will then be applied to Left DLPFC or Left Brodmann Area 6 to investigate cortical excitability changes after ketamine. Electroencephalography(EEG) recordings will be concurrent with TMS procedure.

ASSR/EEG paradigm:

Participants may engage in the auditory steady state response task where click trains of 500-ms duration will be presented binaurally at 65 ± 5 decibel(dB). The click train repetition frequencies will be 40 Hz and presented in the context of an auditory oddball paradigm to ensure participant attention to the stimuli. This task will be done while participants undergo EEG recordings.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18-60 years of age
* Meet criteria for Treatment Resistant Depression (defined as two or more unsuccessful trials of antidepressants at an adequate dose for at least 4 weeks)

Exclusion Criteria:

* Diagnosed with intellectual disability, eg. Mental retardation, neurodegenerative diseases, eg. Early onset neurocognitive disturbances such as frontotemporal dementia or behavioral disorders, eg. adult onset Attention Deficit Hyperactivity Disorder,
* Diagnosed with Bipolar Disorder (BD),
* Diagnosed with personality disorders,
* Previously or currently diagnosed with psychosis (schizoaffective disorder -SAD) or schizophrenia - SCZ),
* Current major medical problems that affect brain anatomy, neurochemistry, or function, e.g., obstructive sleep apnea requiring Continuous Positive Airway Pressure (CPAP), liver insufficiency, kidney insufficiency, cardiovascular problems, systemic infections, cancer, auto-immune diseases, and any brain disorder (seizure disorder, stroke, dementia, degenerative neurologic diseases); history of any brain diseases, including seizures, stroke, meningitis, encephalitis, dementia, degenerative brain diseases, and head injury with loss of consciousness for any period of time,
* Diagnosed specifically with a cardiovascular disorders such as Hypertension, Arrhythmias, Chronic Heart Failure, Myocardial Infarction (MI) or suffering from Chronic Obstructive Pulmonary Disease (COPD) or asthma. Cardiac clearance prior to enrolling in the study and medical records from physician will be required per patient's Primary Care Physician.
* Patients with increased risk of laryngospasm, active upper respiratory infections, respiratory depression, increased intracranial pressure, thyroid disease, or porphyria,
* Current substance abuse or dependence. Only patients who achieved stable, full remission for at least 6 months will be included
* Pregnancy or Breast feeding. All female in reproductive age will undergo pregnancy tests. Female participants will be required to provide evidence of use of contraceptives during the course of the study,
* Unable to understand the design and requirements of the study.
* Unable to sign the informed consent for any reason.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2016-10-14 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2017-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudhakar Selvaraj, MBBS, DPhil, Principal Investigator — University of Texas
Locations (1):
- Harris County Psychiatric Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 subjects signed consent and were screened, but met exclusion criteria and were thus excluded from the study before starting.
  1 subject withdrew consent after screening and did not start the study.
Period: Overall Study
Arm/Group | Ketamine
Started | 5
Completed | 4
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ketamine
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.20 (10.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race data was not collected from 1 participant.
  Participants
    number analyzed (Participants) | 4
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 4
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Cortical Excitability in the Dorsolateral Prefrontal Cortex (DLPFC) as Assessed by Transcranial Magnetic Stimulation-evoked Activity Detected by Electroencephalography (TMS-EEG)
Description: Transcranial magnetic stimulation (TMS) of the left dorsolateral prefrontal cortex (DLPFC) was performed, and electroencephalography (EEG) recording was performed during TMS stimulation. Data is reported as the local mean field amplitude-area under the curve (LMFA-AUC) from a subset of EEG electrodes around the TMS stimulation site.
Time Frame: Baseline
Population: Data was not collected for one participant.
Measure: Mean (Standard Deviation); unit: microvolt * milliseconds (µV * ms)
Arm/Group | Ketamine
Number analyzed (Participants) | 4
microvolt * milliseconds (µV * ms) | 446.08 (209.13)

2. Primary Outcome: Cortical Excitability in DLPFC Using TMS-EEG
Description: as for outcome 1
Time Frame: 4 hours
Population: Data was not collected for 1 participant.
Measure: Mean (Standard Deviation); unit: microvolt * milliseconds (µV * ms)
Arm/Group | Ketamine
Number analyzed (Participants) | 4
microvolt * milliseconds (µV * ms) | 319.71 (206.04)

3. Primary Outcome: Cortical Excitability in DLPFC Using TMS-EEG
Description: as for outcome 1
Time Frame: 24 hours
Population: Data was not collected for 1 participant.
Measure: Mean (Standard Deviation); unit: microvolt * milliseconds (µV * ms)
Arm/Group | Ketamine
Number analyzed (Participants) | 4
microvolt * milliseconds (µV * ms) | 330.30 (222.45)

4. Primary Outcome: Cortical Excitability in DLPFC Using TMS-EEG
Time Frame: 7 days
Population: Data was not collected from any participant at 7 days.
Arm/Group | Ketamine
Number analyzed (Participants) | 0

5. Secondary Outcome: Severity of Depressive Symptoms as Assessed by the Montgomery-Asberg Depression Rating Scale (MADRS)
Description: Total MADRS score ranges from 0 to 60, and a higher score indicates more severe depression, as follows:
  0 to 6 - normal/symptom absent 7 to 19 - mild depression 20 to 34 - moderate depression >34 - severe depression
Time Frame: Baseline
Population: Data was not collected for one participant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine
Number analyzed (Participants) | 4
units on a scale | 24.50 (7.09)

6. Secondary Outcome: Severity of Depressive Symptoms as Assessed by the Montgomery-Asberg Depression Rating Scale (MADRS)
Description: as for outcome 5
Time Frame: 4 hours
Population: Data was not collected for one participant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine
Number analyzed (Participants) | 4
units on a scale | 22.5 (9.73)

7. Secondary Outcome: Severity of Depressive Symptoms as Assessed by the Montgomery-Asberg Depression Rating Scale (MADRS)
Description: as for outcome 5
Time Frame: 24 hours
Population: Data was not collected for one participant.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine
Number analyzed (Participants) | 4
units on a scale | 16.25 (7.66)

8. Secondary Outcome: Safety as Indicated by Number of Adverse Events
Time Frame: 24 hours
Measure: Number; unit: adverse events
Arm/Group | Ketamine
Number analyzed (Participants) | 5
adverse events | 1

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Ketamine
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=5)
Depersonalization (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-02): https://cdn.clinicaltrials.gov/large-docs/95/NCT02935595/Prot_SAP_000.pdf